CLINICAL TRIAL: NCT00933855
Title: A Feasibility Study of a Patient Communication Training Intervention
Brief Title: Patient Communication Training Intervention
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Queens Health Network (Other)
Responsible Party: Sponsor
Other Study IDs: 08-148
Record Dates: First submitted 2009-07-01; First posted 2009-07-07 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Cancer
Keywords: Training Workshop; Communication; Questionnaires; Multiple Diseases
MeSH Terms: conditions — Neoplasms; Communication | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- communication training workshop: The patient intervention is a 1 hour communication workshop entitled: "Getting the Most out of your Doctor's Visit." The workshops will be offered to both patients and family members, but data will be collected only for patients. The workshops will be held on location at Queens Cancer Center.
  Interventions: Behavioral: Questionnaires and training workshop

INTERVENTIONS:
Behavioral: Questionnaires and training workshop — We will recruit a minimum of 1 and maximum of 12 patients for each workshop.
  The workshop will follow the approximate time table below:
  10 minutes: Sign-in, welcome and introductions 25 minutes: Didactic session, videos and discussion 10 minutes: Group discussion 15 minutes: Closing plenary and final assessment

SUMMARY:
The purpose of this study is to test a class for Queens Cancer Center patients. We want to find out if patients think this program is helpful.

DETAILED DESCRIPTION:
It is well accepted that effective physician-patient communication is associated with important outcomes. Communication training interventions for oncologists and other clinicians has been shown to be effective in changing behavior and improving outcomes. Less attention has been given to improving cancer patients' communication with their physicians. Most of the studies in this area have been focused on activating patients through training them to ask questions. Although question asking is a vitally important patient communication skill, other patient communication skills should also be encouraged for patients.

In the primary care setting, studies on patient communication training have focused on three additional communication skills to asking questions: presenting information, checking understanding, and expressing concerns. The goal of this study is to pilot test a patient communication workshop that builds on the work done in the primary care setting, offering an intervention that focuses on a broad range of skills. The proposal aims to improve communication skills in an underserved population, which may be a factor contributing to minority health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeing a physician at Queens Cancer Center (not family members or partners)
* Able to provide informed consent.

Exclusion Criteria:

* Less than 18 years of age (as per self-report)
* Cognitive or physical impairment rendering patients incapable of providing informed consent to participate in the study.
* As the workshop will be given in English and the measures are all written in English, subjects who are not fluent in English will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Queen Cancer Center Clinic waiting room.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of a patient communication training intervention. | 2 years

SECONDARY OUTCOMES:
To attain preliminary data on the acceptability of the intervention through patient ratings of effectiveness and usefulness of the intervention. | 2 years
To attain preliminary data on the effect of a patient communication training intervention on patients' self-reported communication behaviors. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carma Bylund-Lincoln, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Queens Hospital Center, Jamaica, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org